CLINICAL TRIAL: NCT05513391
Title: Immunogenicity and Safety of Quadrivalent Recombinant Influenza Vaccine Compared With Egg-Based Standard-Dose Quadrivalent Influenza Vaccine in Children 3 to 8 Years of Age.
Brief Title: Study With Quadrivalent Recombinant Influenza Vaccine (RIV4) Compared With Egg-Based Quadrivalent Influenza Vaccine (IIV4) in Participants Aged 3 to 8 Years
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to prematurely stop the study. This decision was made without any safety concerns.
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VAP00026; U1111-1256-8841 (Registry Identifier: ICTRP); VAP00026 (Other: Sanofi Identifier); 2022-000576-19 (EudraCT Number)
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Results first posted 2024-07-24 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Influenza Immunization
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Modified double-blind (participant, Sponsor, and Investigator blinded)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- RIV4 cohort (Experimental): RIV4 single injection at Day 1
  Interventions: Biological: Recombinant influenza vaccine (RIV4)
- IIV4 cohort (Active Comparator): IIV4, single injection at Day 1
  Interventions: Biological: Quadrivalent influenza vaccine (IIV4)

INTERVENTIONS:
Biological: Recombinant influenza vaccine (RIV4) — Pharmaceutical form: solution for injection Route of administration: intramuscular
  Other Names: Supemtek / Flublok Quadrivalent
  Arms: RIV4 cohort
Biological: Quadrivalent influenza vaccine (IIV4) — Pharmaceutical form: suspension for injection Route of administration: intramuscular
  Other Names: Fluarix Tetra / Fluarix® Quadrivalent
  Arms: IIV4 cohort

SUMMARY:
The purpose of this study was to demonstrate the non-inferior HAI immune response of quadrivalent recombinant influenza vaccine (RIV4) vs licensed Egg-Based Quadrivalent Influenza Vaccine (IIV4) for the 4 strains based on the egg-derived antigen in all participants aged 3 to 8 years and to describe the immunogenicity and safety profile of RIV4 compared to IIV4 in participants aged 3 to 8 years.

DETAILED DESCRIPTION:
Participants were enrolled on the day of their first vaccination and received 1 or 2 doses 28 days apart of either RIV4 or IIV4; depending on if they were previously vaccinated against influenza or previously unvaccinated against influenza, respectively; and were followed for 6 months after the last vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3 to 8 years on the day of inclusion
* Assent form has been signed and dated by the participant (according to local regulations), and informed consent form has been signed and dated by the parent(s) or another legally acceptable representative and by an independent witness, if required by local regulations

Exclusion Criteria:

* Known or suspected congenital or acquired immunodeficiency, or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* Thrombocytopenia
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination based on the Investigator's judgment
* Personal or family history of Guillain-Barre Syndrome (GBS)
* Personal history of clinically significant development delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder NOTE: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 366 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (31):
- United States (18):
  - Birmingham Pediatric Associates Site Number : 8400023, Birmingham, Alabama
  - The Children's Clinic Of Jonesboro PA Site Number : 8400025, Jonesboro, Arkansas
  - California Research Foundation Site Number : 8400003, San Diego, California
  - Meridian Clinical Research- Sioux City Site Number : 8400007, Sioux City, Iowa
  - AMR - Newton Site Number : 8400021, Newton, Kansas
  - Kentucky Pediatrics / Adult Research Site Number : 8400010, Bardstown, Kentucky
  - Velocity Clinical Research- New Orleans Site Number : 8400012, New Orleans, Louisiana
  - Velocity Clinical Research Lincoln Site Number : 8400013, Lincoln, Nebraska
  - Velocity Clinical Research Omaha Site Number : 8400009, Omaha, Nebraska
  - Meridian Clinical Research Site Number : 8400006, Binghamton, New York
  - Velocity Clinical Research Vestal Site Number : 8400016, Vestal, New York
  - Ohio Pediatric Research Site Number : 8400020, Dayton, Ohio
  - Rainbow Pediatrics Site Number : 8400014, Barnwell, South Carolina
  - Coastal Pediatric Research Charleston Site Number : 8400005, Charleston, South Carolina
  - Coastal Carolina Research Center Site Number : 8400022, North Charleston, South Carolina
  - JBR Clinical Research Site Number : 8400001, Salt Lake City, Utah
  - J. Lewis Research Site Number : 8400017, Salt Lake City, Utah
  - Alliance for Multispecialty Research Syracuse Site Number : 8400027, Syracuse, Utah
- Poland (7):
  - Investigational Site Number : 6160010, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number : 6160007, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number : 6160005, Siemianowice Śląskie, Silesian Voivodeship
  - Investigational Site Number : 6160003, Bydgoszcz
  - Investigational Site Number : 6160006, Tarnów
  - Investigational Site Number : 6160001, Warsaw
  - Investigational Site Number : 6160012, Wroclaw
- Spain (6):
  - Investigational Site Number : 7240014, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240004, Madrid
  - Investigational Site Number : 7240018, Madrid
  - Investigational Site Number : 7240005, Málaga
  - Investigational Site Number : 7240001, Móstoles
  - Investigational Site Number : 7240007, Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VAP00026 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25370&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 31 investigational sites in 3 countries between 10 November 2022 to 03 October 2023.
Pre-assignment Details: A total of 366 participants were enrolled in this study and randomized in a 1:1 ratio to receive quadrivalent recombinant influenza vaccine (RIV4) or quadrivalent inactivated influenza vaccine (IIV4). These participants were stratified according to their previous influenza vaccination status and their age.
Groups:
- RIV4: Participants who were previously vaccinated against influenza received a single intramuscular (IM) injection of RIV4 0.5 milliliter (mL) on Day 1. Participants who were previously unvaccinated against influenza received a single IM injection of RIV4 0.5 mL on Day 1 and Day 29.
- IIV4: Participants who were previously vaccinated against influenza received a single IM injection of IIV4 0.5 mL on Day 1. Participants who were previously unvaccinated against influenza received a single IM injection of IIV4 0.5 mL on Day 1 and Day 29.
Period: Overall Study
Arm/Group | RIV4 | IIV4
Started | 183 | 183
Safety Analysis Set (Safety analysis set included participants who received at least 1 dose of the study vaccine.) | 181 | 181
Completed | 177 | 177
Not Completed | 6 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Deviation | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Withdrawal by Parent/Guardian | 2 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all participants randomized by study interactive response technology to one of the study groups.
Groups:
- RIV4: Participants who were previously vaccinated against influenza received a single IM injection of RIV4 0.5 mL on Day 1. Participants who were previously unvaccinated against influenza received a single IM injection of RIV4 0.5 mL on Day 1 and Day 29.
- Total: Total of all reporting groups
Arm/Group | RIV4 | IIV4 | Total
Number analyzed (Participants) | 183 | 183 | 366
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.73 (1.72) | 5.48 (1.64) | 5.60 (1.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 93 | 188
  Male | 88 | 90 | 178
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 144 | 136 | 280
  Black | 31 | 33 | 64
  American Indian or Alaska Native | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Mixed origin | 4 | 13 | 17
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Influenza Vaccine Antibodies 28 Days After the Last Vaccination
Description: GMTs of influenza vaccine antibodies were measured using individual hemagglutination inhibition (HAI) assay for 4 influenza virus strains: A/H1N1 strain, A/H3N2 strain, B/Victoria lineage strain, and B/Yamagata lineage strain.
Time Frame: Day 29 [participants previously vaccinated] or Day 57 [participants previously unvaccinated]
Population: Analysis was performed on the per-protocol analysis set (PPAS)-subset of full analysis set (FAS) which included participants who received 1 dose of the study vaccine and had a post-vaccination blood sample. Only participants with data collected for each category at Day 29 [participants previously vaccinated] or Day 57 [participants previously unvaccinated] are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | RIV4 | IIV4
Number analyzed (Participants) | 159 | 158
titer
  A/H1N1 | 998 [779 to 1279] | 640 [493 to 831]
  A/H3N2 | 2398 [1914 to 3004] | 889 [722 to 1095]
  B/Victoria | 337 [263 to 432] | 605 [480 to 762]
  B/Yamagata | 789 [634 to 983] | 708 [590 to 850]
Statistical Analysis 1: Comparison: RIV4 vs IIV4; Statistical analysis for A/H1N1; Test type: Non-Inferiority — Non inferiority for GMTs was demonstrated if the lower limit of the 2-sided 95% confidence interval (CI) of the GMT ratio was greater than (>) 0.667 for each virus strain; GMT Ratio = 1.28, 95% CI 2-sided [0.948 to 1.73]
Statistical Analysis 2: Comparison: RIV4 vs IIV4; Statistical analysis for A/H3N2; Test type: Non-Inferiority — Non inferiority for GMTs was demonstrated if the lower limit of the 2-sided 95% CI of the GMT ratio was > 0.667 for each virus strain; GMT Ratio = 2.53, 95% CI 2-sided [1.93 to 3.30]
Statistical Analysis 3: Comparison: RIV4 vs IIV4; Statistical analysis for B/Victoria; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT Ratio = 0.515, 95% CI 2-sided [0.397 to 0.668]
Statistical Analysis 4: Comparison: RIV4 vs IIV4; Statistical analysis for B/Yamagata; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT Ratio = 1.02, 95% CI 2-sided [0.799 to 1.30]

2. Primary Outcome: Percentage of Participants With Seroconversion (SC) Against Antigens 28 Days After the Last Vaccination
Description: Anti-influenza antibodies were measured using HAI assay for 4 influenza virus strains: A/H1N1 strain, A/H3N2 strain, B/Victoria lineage strain, and B/Yamagata lineage strain. SC was defined as either a pre-vaccination HAI titer less than (<) 10 (1/dilution) and a post-vaccination titer greater than or equal to (≥) 40 (1/dilution) or a pre-vaccination titer ≥ 10 (1/dilution) and a ≥ 4-fold increase in post-vaccination titer.
Time Frame: Day 29 [participants previously vaccinated] or Day 57 [participants previously unvaccinated]
Population: Analysis was performed on the PPAS-subset of FAS which included participants who received 1 dose of the study vaccine and had a post-vaccination blood sample. Only participants with data collected for each category at Day 29 [participants previously vaccinated] or Day 57 [participants previously unvaccinated] are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RIV4 | IIV4
Number analyzed (Participants) | 158 | 157
percentage of participants
  A/H1N1 | 84.8 [78.2 to 90.0] | 77.7 [70.4 to 84.0]
  A/H3N2 | 82.3 [75.4 to 87.9] | 66.9 [58.9 to 74.2]
  B/Victoria | 85.4 [79.0 to 90.5] | 92.4 [87.0 to 96.0]
  B/Yamagata | 88.6 [82.6 to 93.1] | 82.8 [76.0 to 88.4]
Statistical Analysis 1: Comparison: RIV4 vs IIV4; Statistical analysis for A/H1N1; Test type: Non-Inferiority — Non-inferiority for SC was demonstrated if the lower limit of the 2-sided 95% CI was > -10% for the 4 strains; Difference in percentage of participants = 7.10, 95% CI 2-sided [-1.55 to 15.7]
Statistical Analysis 2: Comparison: RIV4 vs IIV4; Statistical analysis for A/H3N2; Test type: Non-Inferiority — Non-inferiority for SC was demonstrated if the lower limit of the 2-sided 95% CI was > -10% for the 4 strains; Difference in percentage of participants = 15.4, 95% CI 2-sided [5.80 to 24.7]
Statistical Analysis 3: Comparison: RIV4 vs IIV4; Statistical analysis for B/Victoria; Test type: Non-Inferiority — Non-inferiority for SC was demonstrated if the lower limit of the 2-sided 95% CI was > -10% for the 4 strains; Difference in percentage of participants = -6.91, 95% CI 2-sided [-14.02 to 0.10]
Statistical Analysis 4: Comparison: RIV4 vs IIV4; Statistical analysis for B/Yamagata; Test type: Non-Inferiority — Non-inferiority for SC was demonstrated if the lower limit of the 2-sided 95% CI was > -10% for the 4 strains; Difference in percentage of participants = 5.81, 95% CI 2-sided [-1.99 to 13.6]

3. Secondary Outcome: GMTs of Influenza Vaccine Antibodies at Day 1
Description: GMTs of influenza vaccine antibodies were measured using HAI assay for 4 influenza virus strains: A/H1N1 strain, A/H3N2 strain, B/Victoria lineage strain, and B/Yamagata lineage strain.
Time Frame: Pre-vaccination on Day 1
Population: Analysis was performed on the PPAS-subset of FAS which included participants who received 1 dose of the study vaccine and had a post-vaccination blood sample. Only participants with data collected for each category at Day 1 are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | RIV4 | IIV4
Number analyzed (Participants) | 159 | 157
titer
  A/H1N1 | 70.5 [52.2 to 95.2] | 46.5 [33.9 to 63.7]
  A/H3N2 | 141 [103 to 193] | 112 [81.1 to 156]
  B/Victoria | 20.9 [16.9 to 25.8] | 18.4 [14.9 to 22.7]
  B/Yamagata | 65.2 [50.9 to 83.5] | 54.7 [42.8 to 70.1]

4. Secondary Outcome: Percentage of Participants With Detectable HAI Titer ≥ 10 and ≥ 40 for Influenza Vaccine Antibodies at Day 1 and 28 Days After the Last Vaccination
Description: Antibody titers were measured using HAI assay for 4 influenza virus strains: A/H1N1 strain, A/H3N2 strain, B/Victoria lineage strain, and B/Yamagata lineage strain.
Time Frame: Day 1 (all participants) and Day 29 (participants previously vaccinated) or Day 57 (participants previously unvaccinated)
Population: Analysis was performed on the PPAS-subset of FAS which included participants who received 1 dose of the study vaccine and had a post-vaccination blood sample. Only participants with data collected for each category at Day 1 and Day 29 [participants previously vaccinated] or Day 57 [participants previously unvaccinated] are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RIV4 | IIV4
Number analyzed (Participants) | 159 | 158
percentage of participants
  Titer ≥ 10: A/H1N1: Day 1: number analyzed (Participants) | 159 | 157
  Titer ≥ 10: A/H1N1: Day 1 | 78.6 [71.4 to 84.7] | 70.7 [62.9 to 77.7]
  Titer ≥ 10: A/H1N1: Day 29 or Day 57 | 98.7 [95.5 to 99.8] | 98.1 [94.6 to 99.6]
  Titer ≥ 10: A/H3N2: Day 1: number analyzed (Participants) | 159 | 157
  Titer ≥ 10: A/H3N2: Day 1 | 87.4 [81.2 to 92.1] | 81.5 [74.6 to 87.3]
  Titer ≥ 10: A/H3N2: Day 29 or Day 57 | 100 [97.7 to 100] | 99.4 [96.5 to 100]
  Titer ≥ 10: B/Victoria: Day 1: number analyzed (Participants) | 159 | 157
  Titer ≥ 10: B/Victoria: Day 1 | 69.8 [62.0 to 76.8] | 63.1 [55.0 to 70.6]
  Titer ≥ 10: B/Victoria: Day 29 or Day 57 | 99.4 [96.5 to 100] | 100 [97.7 to 100]
  Titer ≥ 10: B/Yamagata: Day 1: number analyzed (Participants) | 159 | 157
  Titer ≥ 10: B/Yamagata: Day 1 | 85.5 [79.1 to 90.6] | 87.3 [81.0 to 92.0]
  Titer ≥ 10: B/Yamagata: Day 29 or Day 57 | 100 [97.7 to 100] | 100 [97.7 to 100]
  Titer ≥ 40: A/H1N1: Day 1: number analyzed (Participants) | 159 | 157
  Titer ≥ 40: A/H1N1: Day 1 | 65.4 [57.5 to 72.8] | 54.8 [46.6 to 62.7]
  Titer ≥ 40: A/H1N1: Day 29 or Day 57 | 97.5 [93.7 to 99.3] | 96.2 [91.9 to 98.6]
  Titer ≥ 40: A/H3N2: Day 1: number analyzed (Participants) | 159 | 157
  Titer ≥ 40: A/H3N2: Day 1 | 76.1 [68.7 to 82.5] | 70.1 [62.2 to 77.1]
  Titer ≥ 40: A/H3N2: Day 29 or Day 57 | 98.1 [94.6 to 99.6] | 98.1 [94.6 to 99.6]
  Titer ≥ 40: B/Victoria: Day 1: number analyzed (Participants) | 159 | 157
  Titer ≥ 40: B/Victoria: Day 1 | 35.8 [28.4 to 43.8] | 33.8 [26.4 to 41.7]
  Titer ≥ 40: B/Victoria: Day 29 or Day 57 | 92.5 [87.2 to 96.0] | 96.8 [92.8 to 99.0]
  Titer ≥ 40: B/Yamagata: Day 1: number analyzed (Participants) | 159 | 157
  Titer ≥ 40: B/Yamagata: Day 1 | 69.8 [62.0 to 76.8] | 66.2 [58.3 to 73.6]
  Titer ≥ 40: B/Yamagata: Day 29 or Day 57 | 99.4 [96.5 to 100] | 99.4 [96.5 to 100]

5. Secondary Outcome: Geometric Mean Titer Ratio (GMTR) of Influenza Vaccine Antibodies
Description: GMTR was the ratio of the individual titers post-vaccination over pre-vaccination. The GMTs of influenza vaccine antibodies were measured using HAI assay for 4 influenza virus strains: A/H1N1 strain, A/H3N2 strain, B/Victoria lineage strain, and B/Yamagata lineage strain.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | RIV4 | IIV4
Number analyzed (Participants) | 158 | 157
ratio
  A/H1N1 | 14.2 [10.7 to 18.6] | 13.8 [10.2 to 18.8]
  A/H3N2 | 17.1 [12.9 to 22.6] | 7.86 [5.89 to 10.5]
  B/Victoria | 16.0 [12.8 to 20.1] | 32.7 [24.8 to 43.1]
  B/Yamagata | 12.2 [9.96 to 14.9] | 13.1 [10.2 to 16.8]

6. Secondary Outcome: Number of Participants With Immediate Unsolicited Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions, i.e., pre-listed in the case report form (CRF) in terms of diagnosis and onset window post-vaccination. Immediate events were recorded to capture medically relevant unsolicited systemic AEs which occurred within the first 30 minutes after vaccination.
Time Frame: Within 30 minutes post-vaccination on Day 1 (all participants) and Day 29 (participants previously unvaccinated)
Population: Safety analysis set included participants who received at least 1 dose of the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | RIV4 | IIV4
Number analyzed (Participants) | 181 | 181
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Solicited Injection Site Reactions and Systemic Reactions
Description: Solicited injection site reactions were reactions at and around the injection/administration site of the investigational medicinal product (IMP) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRF and considered as being related to the IMP administered at that site. Solicited systemic reactions were systemic AEs observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRF, and those occurring during the specified collection period were always considered related to the IMP even if there was evidence of alternative etiology.
Time Frame: Day 1 to Day 8 (all participants); Day 29 to Day 36 (participants previously unvaccinated)
Population: Safety analysis set included participants who received at least 1 dose of the study vaccine. Only participants with data collected for each category up to 7 days post vaccination are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | RIV4 | IIV4
Number analyzed (Participants) | 179 | 180
Participants
  Solicited injection site reactions | 70 | 76
  Solicited systemic reactions | 50 | 66

8. Secondary Outcome: Number of Participants With Unsolicited AEs
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions, i.e., pre-listed in the CRF in terms of diagnosis and onset window post-vaccination.
Time Frame: Up to Day 29 (all participants); Up to Day 57 (participants previously unvaccinated)
Population: Safety analysis set included participants who received at least 1 dose of the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | RIV4 | IIV4
Number analyzed (Participants) | 181 | 181
Participants | 44 | 47

9. Secondary Outcome: Number of Participants With Medically Attended Adverse Events (MAAEs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An MAAE was a new onset or a worsening of a condition that prompted the participant or participant's parent/legally acceptable representative to seek unplanned medical advice at a physician's office or emergency department.
Time Frame: Up to Day 29 (all participants); Up to Day 57 (participants previously unvaccinated)
Population: Safety analysis set included participants who received at least 1 dose of the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | RIV4 | IIV4
Number analyzed (Participants) | 181 | 181
Participants | 18 | 12

10. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) And Adverse Events of Special Interest (AESI)
Description: An SAE was defined as any adverse event that, at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was other medically important event. An AESI was defined as one of scientific and medical concern specific to the Sponsor's study intervention or program, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor was appropriate.
Time Frame: From the first vaccination up to 6 months after the last vaccination, 209 days
Population: Safety analysis set included participants who received at least 1 dose of the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | RIV4 | IIV4
Number analyzed (Participants) | 181 | 181
Participants
  SAEs | 0 | 1
  AESIs | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first vaccination up to 6 months after the last vaccination, 209 days
Description: Analysis was performed on the safety analysis set.
Arm/Group | RIV4 | IIV4
All-Cause Mortality (participants affected / at risk) | 0/181 | 0/181
Serious Adverse Events (participants affected / at risk) | 0/181 | 1/181
Other Adverse Events (participants affected / at risk) | 86/181 | 98/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIV4 (N=181) | IIV4 (N=181)
Bacterial Infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIV4 (N=181) | IIV4 (N=181)
Chills (General disorders) | 11 (11) | 12 (14)
Injection Site Bruising (General disorders) | 7 (7) | 12 (13)
Injection Site Erythema (General disorders) | 24 (28) | 30 (34)
Injection Site Induration (General disorders) | 17 (18) | 19 (23)
Injection Site Pain (General disorders) | 61 (73) | 66 (76)
Injection Site Swelling (General disorders) | 19 (22) | 17 (18)
Malaise (General disorders) | 35 (37) | 37 (40)
Pyrexia (General disorders) | 12 (13) | 15 (17)
Upper Respiratory Tract Infection (Infections and infestations) | 10 (10) | 11 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 29 (31) | 43 (48)
Headache (Nervous system disorders) | 23 (24) | 32 (35)

LIMITATIONS AND CAVEATS:
Sponsor decision to prematurely stop the study. This decision was made without any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT05513391/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/91/NCT05513391/SAP_001.pdf